CLINICAL TRIAL: NCT04949022
Title: Glycemic Outcomes and Safety With Minimed 780G System in Children With Type 1 Diabetes Aged 2-6 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Medtronic International Trading Sarl (Industry)
Responsible Party: Principal Investigator, Tero Varimo, MD, PhD, MD, PhD, fellow in pediatric endocrinology, principal investigator, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERP-2020-12544
Record Dates: First submitted 2021-06-17; First posted 2021-07-02 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes
Keywords: hybrid closed loop system
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid closed loop system (Experimental): Initiation of 780G insulin pump. First two weeks run-in-phase in open loop Manual mode, followed by a12 month study phase with advanced hybrid closed loop Auto mode.
  Interventions: Device: Medronic 780G insulin pump

INTERVENTIONS:
Device: Medronic 780G insulin pump — Commercial hybrid closed loop system Medronic 780G

SUMMARY:
The purpose of this study is to evaluate the effectiveness of advanced hybrid-closed loop system, Minimed 780G to glycemic control and safety in children aged 2-6 years with type 1 diabetes.

Additionally, the study evaluates the perceived burden of the diabetes treatment to families during the advanced hybrid-closed loop system treatment (diabetes distress).

This is a prospective, non-randomized, single-arm study, where primary endpoint is the change in TIR after hybrid-closed loop system initiation. Secondary endpoints are safety (number of severe hypoglycaemias and diabetic ketoacidosis, DKA), HbA1c, time below range (TBR), mean sensor glucose (SG), standard deviation of SG, and coefficient of variation (CV).

The inclusion criteria are 1) TDD (total insulin daily dose) ≥ 8 units, 2) HbA1c < 10%, 3) capability to use pump and the CGM, and 4) time from diabetes diagnosis more than 6 months. The exclusion criteria are hemophilia or any other bleeding disorder, a condition, which in the opinion of the investigator would put the participant at risk during the trial.

DETAILED DESCRIPTION:
BACKGROUND

The treatment of small children's type 1 diabetes (T1D) is challenging. There is often great day-to-day and within-day variability in glucose levels and HbA1c targets are hard to achieve. The results on hybrid closed loop systems (HCL) in children have been encouraging, suggesting that an algorithm, which automatically doses basal insulin based on sensor glucose (SG) levels, improves time in range (TIR) (3.9-10 mmol/l / 71-180 mg/dl) and reduces the time spent below range (TBR). Despite of these improvements, the target level of TIR (70%) has not been reached in these studies.

In pivotal studies, Minimed 780G advanced HCL system has helped children over 7 years old to reach higher TIR and improve mealtime glycaemia without increasing TBR, severe hypoglycaemias or ketoacidosis.

This study evaluates the effectiveness to glycemic control and safety of advanced hybrid-closed loop system, Minimed 780G, in children aged between 2.0-6.99 years, with type 1 diabetes.

The study protocol is explained to the participants (2.0-6.99 year-old children) orally. Informed consent from participants' caregivers and those participants who can write will be taken by investigators, clinicians or diabetes nurses. The investigator will explain the nature of the study to the subject, and answer all questions regarding this study. Prior to any study-related screening procedures being performed on the participant, the informed consent statement will be reviewed and signed and dated by participant's caregiver.

STUDY PROTOCOL

The study includes a two week run-in-phase in open loop Manual mode, which equals for standard sensor augmented pump (SAP) treatment (this feature is also in the same device), which is followed by a three month study phase with advanced hybrid closed loop Auto mode.

The participants will be given an advanced HCL pump (MiniMed 780G™ system with SmartGuard Medtronic, Northridge, CA). Minimed 780g™ is an insulin pump, which doses insulin automatically to patients subcutaneous tissue every 5 minutes based on SG values. The maximal dosing is based on participants TDD. The SmartGuard feature uses meal information, up to date SG reading, and SG target values to control basal insulin delivery. Additionally, it can automatically deliver a correction bolus to correct a high SG reading. The MiniMed 780G insulin pump requires a minimum of eight units and a maximum of 250 units per day to operate using the SmartGuard feature (Medtronic Minimed 780g™ system user guide).

This device has CE mark and is indicated to children aged over 7 years who require insulin over 8 units/day. In manufacturers safety studies, no adverse effects (diabetic ketoacidosis (DKA) or severe hypoglycaemias) has been reported in children over 7 years old who had TDD over 8 units/day (MDT personal communication).

The infusion set of insulin pump is changed every 2-3 days by patients' caregivers. The material connected to subcutaneous tissue is Teflon. The SG values are measured by continuous glucose monitor (CGM). The used CGM is Guardian3 sensor, which is integrated to Minimed 780g™ system. It measures the glucose level in the subcutaneous tissue. The CGM sensor connects to a transmitter that sends the glucose data to insulin pump. The sensor is worn for 7 days and then replaced with a new one by the participants' caregivers.

The traceability is achieved by each device's serial number (insulin pump, CGM transmitter). The glucose sensors, infusion sets, reservoirs and glucose sensors have lot numbers.

The families are trained to use the device by Medtronic's local representatives (technical issues), diabetes nurses, and clinicians (dosing and other medical issues). If the family has been on a sensor augmented pump (SAP) treatment previously, training includes one 3 hour session, a normal procedure in our clinic, at the outpatient clinic. If family has no previous experience on pump treatment or CGM, they will first try CGM out for 2 weeks and then 3-days visit on day hospital is arranged to first learn the basics on insulin pump treatment.

POWER ANALYSES

Based on previous studies, it was estimated that a significant difference in increased TIR between the advanced HCL treatment and the Manual mode would be 10% and the standard deviation is expected to be 13%. Taken these into account, the power of 90% to detect a difference between the modes with type 1 error rate of 0.05, 35 participants should complete the protocol. The dropout rate is estimated to be less than 3%, thus 38 HCL systems have been reserved for 38 participants.

ETHICAL ISSUES

This study is conducted in accordance with the ethical principles that have their origins in the Declaration of Helsinki. This study will be conducted in accordance with Good Clinical Practice (GCP), as defined by the International Conference on Harmonization (ICH) and in accordance with the ethical principles underlying European Union Directive 2001/20/EC and 2005/28/EC (or Regulation (EU) No 536/2014). The ethics committee of Helsinki University Hospital and The Finnish Medicines Agency has approved the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* total insulin daily dose ≥ 8 units
* HbA1c < 10%
* capability to use pump and the CGM
* time from diabetes diagnosis more than 6 months

Exclusion Criteria:

* hemophilia or any other bleeding disorder, a condition, which in the opinion of the investigator would put the participant at risk during the trial

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time in range (glucose between 3.9-10 mmol/l) before and during hybrid close loop insulin pump treatment | Up to 3 months
  Time in range (%) derived from continuous glucose monitoring
Time in range (glucose between 3.9-10 mmol/l) before and during hybrid close loop insulin pump treatment | Up to 12 months
  Time in range (%) derived from continuous glucose monitoring

SECONDARY OUTCOMES:
The number of severe hypoglycemia before and during hybrid close loop insulin pump treatment | Up to 3 months
  Number of hypoglycemia (glucose <3.0 and altered mental status) derived from blood glucose monitoring
The number of severe hypoglycemia before and during hybrid close loop insulin pump treatment | Up to 12 months
  Number of hypoglycemia (glucose <3.0 and altered mental status) derived from blood glucose monitoring
Number of diabetic ketoacidosis in participant before and during hybrid close loop insulin pump treatment | Up to 3 months
  Number of diabetes ketoacidosis derived from patient information system
Number of diabetic ketoacidosis in participant before and during hybrid close loop insulin pump treatment | Up to 12 months
  Number of diabetes ketoacidosis derived from patient information system
Diabetes distress before and during hybrid close loop insulin pump treatment | Up to 3 months
  Parents diabetes distress measured with validated questionnaire: Problem Areas In Diabetes-Parent Revised (PAID-Pr) (scored 0-72)
Diabetes distress before and during hybrid close loop insulin pump treatment | Up to 12 months
  Parents diabetes distress measured with validated questionnaire: Problem Areas In Diabetes-Parent Revised (PAID-Pr) (scored 0-72)
HbA1c before and during hybrid close loop insulin pump treatment | Up to 3 months
  HbA1c (mmol/mol, %) measured from blood during treatment
HbA1c before and during hybrid close loop insulin pump treatment | Up to 12 months
  HbA1c (mmol/mol, %) measured from blood during treatment

OTHER OUTCOMES:
Time below range (glucose <3.9mmol/l) before and during hybrid close loop insulin pump | Up to 3 months
  Time below range (%) derived from continuous glucose monitoring
Time below range (glucose <3.9mmol/l) before and during hybrid close loop insulin pump | Up to 12 months
  Time below range (%) derived from continuous glucose monitoring
Mean sensor glucose before and during hybrid close loop insulin pump | Up to 3 months
  Mean sensor glucose (mmol/l) derived from continuous glucose monitoring
Mean sensor glucose before and during hybrid close loop insulin pump | Up to 12 months
  Mean sensor glucose (mmol/l) derived from continuous glucose monitoring
Sensor glucose standard deviation before and during hybrid close loop insulin pump | Up to 3 months
  Sensor glucose standard deviation (mmol/l) derived from continuous glucose monitoring
Sensor glucose standard deviation before and during hybrid close loop insulin pump | Up to 12 months
  Sensor glucose standard deviation (mmol/l) derived from continuous glucose monitoring
Sensor glucose coefficient of variation before and during hybrid close loop insulin pump | Up to 3 months
  Sensor glucose coefficient of variation (%) derived from continuous glucose monitoring
Sensor glucose coefficient of variation before and during hybrid close loop insulin pump | Up to 12 months
  Sensor glucose coefficient of variation (%) derived from continuous glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Kaisa Tuomaala, MD, PhD, Principal Investigator — Helsinki University Hospital, New Children's Hospital
Locations (1):
- Helsinki University Hospital, New Children's Hospital and Jorvi Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: 24 months after the completion of the study
Access Criteria: Data will be shared according to the EU General Data Protection Regulation and national and hospital data protection regulations.

REFERENCES:
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Breton MD, Kanapka LG, Beck RW, Ekhlaspour L, Forlenza GP, Cengiz E, Schoelwer M, Ruedy KJ, Jost E, Carria L, Emory E, Hsu LJ, Oliveri M, Kollman CC, Dokken BB, Weinzimer SA, DeBoer MD, Buckingham BA, Chernavvsky D, Wadwa RP; iDCL Trial Research Group. A Randomized Trial of Closed-Loop Control in Children with Type 1 Diabetes. N Engl J Med. 2020 Aug 27;383(9):836-845. doi: 10.1056/NEJMoa2004736. PMID 32846062
- [Background] Lind M, Pivodic A, Svensson AM, Olafsdottir AF, Wedel H, Ludvigsson J. HbA1c level as a risk factor for retinopathy and nephropathy in children and adults with type 1 diabetes: Swedish population based cohort study. BMJ. 2019 Aug 28;366:l4894. doi: 10.1136/bmj.l4894. PMID 31462492
- [Background] Hagger V, Hendrieckx C, Sturt J, Skinner TC, Speight J. Diabetes Distress Among Adolescents with Type 1 Diabetes: a Systematic Review. Curr Diab Rep. 2016 Jan;16(1):9. doi: 10.1007/s11892-015-0694-2. PMID 26748793
- [Derived] Pulkkinen MA, Varimo TJ, Hakonen ET, Harsunen MH, Hyvonen ME, Janer JN, Kiiveri SM, Laakkonen HM, Laakso SM, Wehkalampi K, Hero MT, Miettinen PJ, Tuomaala AK. MiniMed 780G in 2- to 6-Year-Old Children: Safety and Clinical Outcomes After the First 12 Weeks. Diabetes Technol Ther. 2023 Feb;25(2):100-107. doi: 10.1089/dia.2022.0313. Epub 2022 Dec 30. PMID 36511831